CLINICAL TRIAL: NCT01021618
Title: The Ex-Lex Trial: A Randomized Trial Combining Regadenoson With Symptom-Limited Exercise in Patients Undergoing Myocardial Perfusion Imaging
Brief Title: Regadenoson Combined With Symptom-Limited Exercise in Patients Undergoing Myocardial Perfusion Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HELL002965HI
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — regadenoson; Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vasodilator-exercise stress (Active Comparator): Four-minute infusion of dipyridamole (0.56 mg/kg) followed by symptom-limited exercise; injection of technetium-99m labeled radiopharmaceutical at peak hyperemia or peak exercise followed by SPECT myocardial perfusion imaging
  Interventions: Other: Symptom-limited exercise
- Exercise-vasodilator stress (Experimental): Symptom-limited exercise followed by a bolus intravenous injection of regadenoson (0.4 mg/5 mL) in patients failing to achieve a standard clinical endpoint; injection of technetium-99m labeled radiopharmaceutical 15 seconds after administration of regadenoson (or at peak exercise if regadenoson not administered) followed by SPECT myocardial perfusion imaging.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Regadenoson (0.4mg/5 mL) injection during symptom-limited exercise with technetium-99m SPECT myocardial perfusion imaging
  Other Names: Lexiscan; Exercise-lexiscan stress test
  Arms: Exercise-vasodilator stress
Other: Symptom-limited exercise — Dipyridamole (0.56 mg/kg) over 4 minutes followed by symptom-limited exercise with technetium-99m SPECT myocardial perfusion imaging
  Other Names: Persantine; Persantine-exercise stress test
  Arms: Vasodilator-exercise stress

SUMMARY:
Not infrequently, a physician is faced with uncertainty regarding the ability of a patient to perform adequate exercise in the noninvasive evaluation of known or suspected coronary artery disease (CAD) by the use of radionuclide stress myocardial perfusion imaging. In selected patients, protocols that combine exercise (either low-level or symptom-limited) with vasodilator stress agents have been found to be safe and effective in both identification of the presence and severity of CAD as well as risk stratification for adverse cardiac outcome. However, currently utilized combined stress protocols have drawbacks. Further refinement of combined stress protocols would potentially lead to more appropriate stress protocol selection for patients while enhancing laboratory efficiency. The purpose of this prospective, randomized study will be to evaluate the relative merits of combining regadenoson with symptom-limited exercise in patients clinically-referred for vasodilator-exercise stress myocardial perfusion imaging for the assessment of known or suspected CAD. It is hypothesized that combining regadenoson with symptom-limited exercise is a safe and feasible stress testing modality which is non-inferior to that which combines symptom-limited exercise with dipyridamole.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-nursing females clinically referred for vasodilator stress myocardial perfusion imaging with the addition of exercise
* Age >=30 years

Exclusion Criteria:

* Extremely limited functional capacity
* Age <30 years
* Unable or unwilling to provide informed consent
* Pregnant or nursing females
* Current use of methylxanthines within 12 hours of testing
* Current use of dipyridamole or aminophylline within 48 hours of testing
* Uncontrolled hypertension (>200 mmHg systolic/>120 mmHg diastolic)
* Known hypertrophic cardiomyopathy with obstruction or severe aortic stenosis
* Decompensated congestive heart failure
* History of sick sinus syndrome or > first degree atrioventricular block in the absence of a functioning pacemaker
* Asthma or other bronchospastic reactive airway disease
* History of percutaneous coronary intervention or coronary artery bypass grafting, or documented history of acute myocardial infarction or unstable angina within one week of testing
* Patients at risk for hypotensive reaction to regadenoson

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary V Heller, MD, PhD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Ignaszewski AP, McCormick LX, Heslip PG, McEwan AJ, Humen DP. Safety and clinical utility of combined intravenous dipyridamole/symptom-limited exercise stress test with thallium-201 imaging in patients with known or suspected coronary artery disease. J Nucl Med. 1993 Dec;34(12):2053-61. PMID 8254386
- [Background] Ahlberg AW, Baghdasarian SB, Athar H, Thompsen JP, Katten DM, Noble GL, Mamkin I, Shah AR, Leka IA, Heller GV. Symptom-limited exercise combined with dipyridamole stress: prognostic value in assessment of known or suspected coronary artery disease by use of gated SPECT imaging. J Nucl Cardiol. 2008 Jan-Feb;15(1):42-56. doi: 10.1016/j.nuclcard.2007.09.025. PMID 18242479
- [Background] Thomas GS, Thompson RC, Miyamoto MI, Ip TK, Rice DL, Milikien D, Lieu HD, Mathur VS. The RegEx trial: a randomized, double-blind, placebo- and active-controlled pilot study combining regadenoson, a selective A(2A) adenosine agonist, with low-level exercise, in patients undergoing myocardial perfusion imaging. J Nucl Cardiol. 2009 Jan-Feb;16(1):63-72. doi: 10.1007/s12350-008-9001-9. Epub 2009 Jan 20. PMID 19152130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in the Hartford Hospital Nuclear Cardiology Laboratory from January 2010 and February 2012.
Pre-assignment Details: At the onset of the study, only subjects with scores greater than or equal to 9.95 were randomized. After the first 96 patients had been screened and 55 randomized with no adverse events in the study group, this restriction was removed.
Groups:
- Vasodilator-exercise Stress: Four-minute infusion of dipyridamole (0.56 mg/kg) followed by symptom-limited exercise.
- Exercise-vasodilator Stress: Symptom-limited exercise followed by a bolus intravenous injection of regadenoson (0.4 mg/5 mL) only in patients failing to achieve a standard clinical endpoint
Period: Overall Study
Arm/Group | Vasodilator-exercise Stress | Exercise-vasodilator Stress
Started | 44 | 96
Completed | 44 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasodilator-exercise Stress | Exercise-vasodilator Stress | Total
Number analyzed (Participants) | 44 | 96 | 140
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 63 (11) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 44 | 67
  Male | 21 | 52 | 73
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 21 | 50 | 71
  Hispanic | 13 | 24 | 37
  Black | 8 | 19 | 27
  Other | 2 | 3 | 5
Known Coronary Artery Disease [Number; unit: participants] — History of either myocardial infarction or coronary revascularization
  participants
    Any known coronary disease | 15 | 29 | 44
    No known coronary disease | 29 | 67 | 96
Indication for Stress Testing [Number; unit: participants] — Clinical indication for referral to the nuclear laboratory for stress testing, from the referring clinician
  participants
    Chest Pain | 36 | 71 | 107
    Dyspnea | 4 | 8 | 12
    Arrhythmia | 1 | 7 | 8
    Syncope or Near-Syncope | 2 | 4 | 6
    Other | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events or Side Effects Graded "Severe" on Symptom Questionnaire
Description: Number of participants with any side effect (flushing, shortness of breath, headache, chest discomfort, dizziness, nausea, or abdominal pain) requiring specific treatment or graded as "severe" by the patient; or any death, myocardial infarction, or unplanned hospitalization. Note that 2 patients allocated to exercise-vasodilator stress did not complete symptom questionnaires and are therefore excluded from analysis.
Time Frame: 24 hours
Population: Note that 2 patients allocated to exercise-vasodilator stress did not complete symptom questionnaires and are therefore excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Vasodilator-exercise Stress | Exercise-vasodilator Stress
Number analyzed (Participants) | 44 | 94
participants | 11 | 15

2. Secondary Outcome: Myocardial Perfusion Image Quality
Description: Single photon emission computed tomography myocardial perfusion acquisition and image processing was performed in accordance with American Society of Nuclear Cardiology guidelines. All images were interpreted by consensus read of three investigators blinded to stress test protocol and results. Overall perfusion and gated image quality were described as excellent (no artifacts interfering with myocardial perfusion interpretation), good, fair, or poor (artifact requiring reprocessing or repeat imaging of the patient to allow for diagnostic interpretation).
Time Frame: 0 hours
Population: Note that images were unavailable in one vasodilator-exercise patient because of urgent catheterization after stress test without imaging and one exercise-vasodilator patient for technical reasons.
Measure: Number; unit: participants
Arm/Group | Vasodilator-exercise Stress | Exercise-vasodilator Stress
Number analyzed (Participants) | 43 | 95
participants
  Excellent | 13 | 33
  Good | 25 | 55
  Fair | 5 | 7
  Poor | 0 | 0

ADVERSE EVENTS:
Description: Note that 2 patients allocated to exercise-vasodilator stress did not complete symptom questionnaires and were excluded from the "other adverse events" analysis.
Arm/Group | Vasodilator-exercise Stress | Exercise-vasodilator Stress
Serious Adverse Events (participants affected / at risk) | 2/44 | 2/96
Other Adverse Events (participants affected / at risk) | 11/44 | 14/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vasodilator-exercise Stress (N=44) | Exercise-vasodilator Stress (N=96)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (General disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vasodilator-exercise Stress (N=44) | Exercise-vasodilator Stress (N=94)
Severe Flushing (General disorders) | 2 (2) | 1 (1)
Severe Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (13)
Severe Headache (Nervous system disorders) | 3 (3) | 0 (0)
Severe Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Severe Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Severe Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Severe Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes